CLINICAL TRIAL: NCT04889118
Title: A Phase 3 Randomized, Placebo-controlled Trial to Evaluate the Safety and Efficacy of Pembrolizumab (MK-3475) and Lenvatinib (E7080/MK-7902) Versus Pembrolizumab Alone as First-line Intervention in Participants With Advanced Melanoma (LEAP-003)
Brief Title: Safety and Efficacy Study of Pembrolizumab (MK-3475) Combined With Lenvatinib (MK-7902/E7080) as First-line Intervention in Adults With Advanced Melanoma (MK-7902-003/E7080-G000-312/LEAP-003)-China Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7902-003 China Extension; MK-7902-003 (Other: MSD Protocol Number); E7080-G000-312 (Other: Eisai Protocol Number); LEAP-003 (Other: MSD)
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Malignant Melanoma
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death-ligand 1 (PD-L1, PDL1); programmed cell death-ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+Lenvatinib (Experimental): Participants receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule daily for up to at least 2 years.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- Pembrolizumab+Placebo (Active Comparator): Participants receive pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule daily for up to at least 2 years.
  Interventions: Biological: Pembrolizumab; Drug: Placebo for lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Lenvatinib — Oral capsule
  Other Names: MK-7902; E7080; LENVIMA®
  Arms: Pembrolizumab+Lenvatinib
Drug: Placebo for lenvatinib — Oral capsule
  Arms: Pembrolizumab+Placebo

SUMMARY:
The purpose of the China Extension study is to assess the safety and efficacy of pembrolizumab (MK-3475) combined with lenvatinib (MK-7902/E7080) compared to pembrolizumab alone (with placebo for lenvatinib) as first-line treatment in Chinese participants with no prior systemic therapy for their advanced melanoma.

DETAILED DESCRIPTION:
As of 03-Apr-2023, active participants, investigator, and sponsor personnel or delegate(s) involved in the treatment administration or clinical evaluation of the participants will be unblinded.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed melanoma.
* Has unresectable Stage III or Stage IV melanoma, as per American Joint Committee on Cancer guidelines, not amenable to local therapy.
* Has been untreated for advanced or metastatic disease except as follows: a. proto-oncogene B-Raf (BRAF) V600 mutation-positive melanoma may have received standard of care targeted therapy as first-line therapy for advanced or metastatic disease. Participants that do not have a BRAF V600 mutation but did receive BRAF or BRAF/MEKi therapy are eligible to participate in this study after discussion with the medical monitor.

  b. Prior adjuvant or neoadjuvant therapy, with targeted therapy or immunotherapy (such as anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], anti-programmed cell death 1 [anti-PD-1] therapy or interferon) will only be permitted if relapse did not occur during active treatment or within 6 months of treatment discontinuation.
* Have documentation of BRAF V600-activating mutation status or consent to BRAF V600 mutation testing during the Screening period (participants with BRAF mutation-positive melanoma as well as BRAF wild-type or unknown are eligible).
* Has an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Has the presence of ≥1 measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1.
* Provides a tumor biopsy. Participants must submit tumor sample during Screening for confirmation of adequacy of tumor tissue at a central pathology laboratory. Participants who do not submit a tumor tissue sample will not be randomized. The tumor biopsy may not be obtained from a lone target lesion. Confirmation of presence of tumor tissue is not required prior to randomization.
* Has resolution of toxic effect(s) of the most recent prior therapy to Grade 1 or less (except alopecia). If participant received major surgery or radiation therapy of >30 Gray (Gy), they must have recovered from the toxicity and/or complications from the intervention.
* Male participants must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants must not be pregnant, not breastfeeding, and ≥1 of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to use study-approved contraception during the treatment period and for at least 120 days after the last dose of study treatment.
* The participant (or legally acceptable representative) has provided documented informed consent for the study.
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mmHg at screening and no change in antihypertensive medications within 1 week before Cycle 1 Day 1.
* Has adequate organ function.

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment.
* Has a known additional malignancy that is progressing or requires active treatment.

Exceptions include early stage cancers (carcinoma in situ or Stage 1, non-ulcerated primary melanoma <1 mm in depth with no nodal involvement) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy.

* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has ocular melanoma.
* Has known hypersensitivity to active substances or any of their excipients including previous clinically significant hypersensitivity reaction to treatment with another monoclonal antibody.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has an active infection requiring systemic therapy.
* Has known history of human immunodeficiency virus (HIV) infection.
* Has known history of or is positive for hepatitis B virus or hepatitis C virus infection.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a history of active tuberculosis (Bacillus tuberculosis).
* Has presence of gastrointestinal condition including malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
* Has had a major surgery within 4 weeks prior to Cycle 1 Day 1. Adequate wound healing after major surgery must be assessed clinically and have resolved completely prior to Cycle 1 Day 1.
* Has a pre-existing Grade ≥3 gastrointestinal or non-gastrointestinal fistula.
* Has radiographic evidence of major blood vessel invasion/infiltration.
* Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study treatment.
* Has clinically significant cardiovascular disease within 12 months of the first dose of study treatment including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.
* Has urine protein ≥1 g/24-hour. Note: Participants with ≥2+ (≥100 mg/dL) proteinuria on urine dipstick testing (or urinalysis) will undergo 24-hour urine collection for quantitative assessment of proteinuria.
* Prolongation of QTcF interval to >480 ms. Note: If the QTcF is prolonged to >480 ms in the presence of a pacemaker, contact the Sponsor to determine eligibility.
* Has left ventricular ejection fraction (LVEF) below the institutional (or local laboratory) normal range, as determined by multigated acquisition scan (MUGA) or echocardiogram.
* Has received prior therapy in the adjuvant setting. Note: Targeted therapy, anti-CTLA-4, or anti-PD-1 may be allowed.
* Has received prior systemic treatment for unresectable or metastatic melanoma other than targeted therapy as noted in Inclusion Criteria above.
* Has received prior therapy with a monoclonal antibody, chemotherapy, or an investigational agent or device within 4 weeks or 5 half-lives (whichever is longer) before administration of study treatment or not recovered (≤Grade 1 or at Baseline) from adverse events due to previously administered agents.

Exception to this rule would be use of denosumab, which is not excluded. Note: Participants with alopecia and ≤Grade 2 neuropathy are an exception and may enroll.

* Has received prior radiotherapy within 2 weeks of first dose of study treatment (Cycle 1 Day 1). Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Has received live vaccine within 30 days before the first dose of study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has had an allogeneic tissue/solid organ transplant.
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (11):
- China (11):
  - Beijing Cancer Hospital (0601), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0612), Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center (0602), Guangzhou, Guangdong
  - Henan Cancer Hospital ( Site 0610), Zhengzhou, Henan
  - Nanjing Drum Tower Hospital (0609), Nanjing, Jiangsu
  - The First Hospital Of Jilin University (0603), Changchun, Jilin
  - Fudan University Shanghai Cancer Center ( Site 0607), Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital (0606), Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital (0604), Kunming, Yunnan
  - Sir Run Run Shaw Hospital (0605), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0608), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The China extension study enrolled 131 participants. 62 participants were randomized in the global portion for MK-7902-003 (NCT03820986) and 69 in the China extension portion
Groups:
- Pembrolizumab+Lenvatinib: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule daily for up to at least 2 years.
- Pembrolizumab+Placebo: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule daily for up to at least 2 years.
Period: Overall Study
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Started | 64 | 67
Completed | 0 | 0
Not Completed | 64 | 67
Not completed — Death | 49 | 47
Not completed — Sponsor Decision | 15 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo | Total
Number analyzed (Participants) | 64 | 67 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.4 (11.7) | 57.3 (13.5) | 56.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 32 | 58
  Male | 38 | 35 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 61 | 66 | 127
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 64 | 67 | 131
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) Per Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS is defined as the time from date of randomization to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD. For this study, RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to approximately 30 months
Population: All randomized China participants, included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 64 | 67
Months | 6.1 [4.1 to 8.1] | 2.0 [2.0 to 2.1]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Pembrolizumab+Placebo; Test type: Superiority — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; p = 0.0013, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.37 to 0.81] — HR=Pembrolizumab + Lenvatinib vs. Pembrolizumab + Placebo

2. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to date of death from any cause.
Time Frame: Up to approximately 30 months
Population: All randomized China participants, included in the treatment group to which they were randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 64 | 67
Months | 19.9 [11.9 to 26.8] | 17.0 [12.7 to 25.7]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Pembrolizumab+Placebo; Test type: Superiority — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; p = 0.3728, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.58 to 1.48] — HR=Pembrolizumab + Lenvatinib vs. Pembrolizumab + Placebo

3. Secondary Outcome: Objective Response Rate (ORR) as Assessed by BICR Per RECIST 1.1
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. For this study, RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to approximately 30 months
Population: All randomized China participants, included in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 64 | 67
Percentage of Participants | 26.6 [16.3 to 39.1] | 16.4 [8.5 to 27.5]

4. Secondary Outcome: Duration of Response (DOR) as Assessed by BICR Per RECIST 1.1
Description: For participants who demonstrated CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), DOR is defined as the date of the first documented evidence of CR or PR until PD or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD. For this study, RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to approximately 30 months
Population: Randomized participants who had a confirmed complete or partial response, included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 17 | 11
Months | 13.7 [4.2 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse | NA [6.5 to NA] — NA = Median, upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to approximately 50 months
Population: All randomized participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 64 | 67
Participants | 64 | 67

6. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to Adverse Events (AEs)
Description: The number of participants who discontinue study treatment due to an AE will be presented.
Time Frame: Up to approximately 39 months
Population: All randomized participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 64 | 67
Participants | 10 | 3

ADVERSE EVENTS:
Time Frame: Up to approximately 51 months
Description: The population for all-cause mortality includes all participants in the treatment arm to which they were randomized. The population for SAE and other AEs includes all randomized participants who received at least 1 dose of study intervention. Per protocol, MedDRA V25.1 preferred terms 'Neoplasm progression' , 'Malignant neoplasm progression' and 'Disease progression' not related to the drug are excluded.
Groups:
- Pembrolizumab + Placebo: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule daily for up to at least 2 years.
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab + Placebo
All-Cause Mortality (participants affected / at risk) | 49/64 | 47/67
Serious Adverse Events (participants affected / at risk) | 14/64 | 12/67
Other Adverse Events (participants affected / at risk) | 64/64 | 66/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Lenvatinib (N=64) | Pembrolizumab + Placebo (N=67)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Immune-mediated encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Lenvatinib (N=64) | Pembrolizumab + Placebo (N=67)
Anaemia (Blood and lymphatic system disorders) | 15 (22) | 19 (25)
Hyperthyroidism (Endocrine disorders) | 10 (10) | 11 (13)
Hypothyroidism (Endocrine disorders) | 47 (86) | 15 (16)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8) | 2 (3)
Constipation (Gastrointestinal disorders) | 5 (7) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 26 (37) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 5 (5) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 4 (4) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 7 (10) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 7 (7)
Toothache (Gastrointestinal disorders) | 8 (10) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (14) | 0 (0)
Asthenia (General disorders) | 4 (4) | 4 (4)
Pyrexia (General disorders) | 6 (8) | 4 (6)
COVID-19 (Infections and infestations) | 7 (8) | 8 (8)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 5 (11) | 10 (11)
Alanine aminotransferase increased (Investigations) | 25 (40) | 22 (29)
Amylase increased (Investigations) | 5 (6) | 6 (10)
Aspartate aminotransferase increased (Investigations) | 30 (45) | 17 (19)
Bilirubin conjugated increased (Investigations) | 7 (16) | 8 (17)
Blood alkaline phosphatase increased (Investigations) | 6 (9) | 5 (15)
Blood bilirubin increased (Investigations) | 16 (28) | 16 (36)
Blood bilirubin unconjugated increased (Investigations) | 6 (12) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 10 (10) | 14 (20)
Blood creatinine increased (Investigations) | 9 (16) | 7 (15)
Blood glucose increased (Investigations) | 9 (9) | 5 (6)
Blood lactate dehydrogenase increased (Investigations) | 28 (65) | 17 (23)
Blood thyroid stimulating hormone increased (Investigations) | 10 (13) | 3 (3)
Blood urea increased (Investigations) | 10 (14) | 7 (18)
C-reactive protein increased (Investigations) | 7 (20) | 11 (20)
Electrocardiogram ST-T change (Investigations) | 5 (5) | 7 (8)
Gamma-glutamyltransferase increased (Investigations) | 26 (50) | 18 (24)
Lipase increased (Investigations) | 15 (24) | 4 (4)
Lymphocyte count decreased (Investigations) | 4 (11) | 2 (2)
Neutrophil count decreased (Investigations) | 11 (36) | 4 (4)
Platelet count decreased (Investigations) | 14 (23) | 3 (5)
Red blood cells urine positive (Investigations) | 8 (14) | 5 (7)
Serum amyloid A protein increased (Investigations) | 6 (13) | 9 (12)
Urinary occult blood positive (Investigations) | 10 (18) | 12 (24)
Urobilinogen urine increased (Investigations) | 4 (4) | 0 (0)
Weight decreased (Investigations) | 36 (49) | 15 (18)
White blood cell count decreased (Investigations) | 12 (33) | 5 (10)
White blood cells urine positive (Investigations) | 12 (34) | 7 (19)
Decreased appetite (Metabolism and nutrition disorders) | 18 (20) | 11 (11)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 33 (75) | 13 (28)
Hyperglycaemia (Metabolism and nutrition disorders) | 27 (53) | 9 (17)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 42 (111) | 25 (46)
Hyperuricaemia (Metabolism and nutrition disorders) | 26 (51) | 15 (26)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 (35) | 11 (16)
Hypocalcaemia (Metabolism and nutrition disorders) | 11 (16) | 4 (7)
Hypochloraemia (Metabolism and nutrition disorders) | 7 (7) | 6 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (21) | 8 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (19) | 11 (14)
Hypoproteinaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4) | 4 (5)
Headache (Nervous system disorders) | 5 (6) | 2 (2)
Haematuria (Renal and urinary disorders) | 6 (10) | 5 (6)
Proteinuria (Renal and urinary disorders) | 46 (103) | 31 (58)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Leukoderma (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 18 (20) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (11)
Rash (Skin and subcutaneous tissue disorders) | 11 (14) | 8 (8)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Hypertension (Vascular disorders) | 41 (57) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT04889118/Prot_SAP_002.pdf